CLINICAL TRIAL: NCT03932435
Title: A Open-Label, Randomized, 2-sequence, 2-period, Fasted Condition, Single-dose, Per Oral, Cross-over Study to Evaluate the Bioequivalence of "Dong-a Bepotastine Besilate Tab" (Bepotastine Besilate 10mg) and "Twolion Tab" (Bepotastine Besilate 10mg) in Healthy Volunteers
Brief Title: Bioequivalence Test of "Dong-a Bepotastine Besilate Tab" and "Twolion Tab"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TWLO_BE_01
Record Dates: First submitted 2019-04-22; First posted 2019-04-30 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: single-dose, 2-sequence
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TWLO_C → TWLO (Experimental): TWLO_C: "Dong-a Bepotastine Besilate Tab" (Bepotastine Besilate 10mg), TWLO: "Twolion Tab" (Bepotastine Besilate 10mg)
  Interventions: Drug: Fisrt period TWLO_C; Other: Washout period; Drug: Second period TWLO
- TWLO → TWLO_C (Experimental): TWLO_C: "Dong-a Bepotastine Besilate Tab" (Bepotastine Besilate 10mg), TWLO: "Twolion Tab" (Bepotastine Besilate 10mg)
  Interventions: Drug: Fisrt period TWLO; Other: Washout period; Drug: Second period TWLO_C

INTERVENTIONS:
Drug: Fisrt period TWLO_C — First Period: Single oral administration of 1 tablet of "Dong-a Bepotastine Besilate Tab"(Bepotastine Besilate 10mg)
  Other Names: "Dong-a Bepotastine Besilate Tab"
  Arms: TWLO_C → TWLO
Drug: Fisrt period TWLO — First Period: Single oral administration of 1 tablet of "Twolion Tab"(Bepotastine Besilate 10mg)
  Other Names: "Twolion Tab"
  Arms: TWLO → TWLO_C
Other: Washout period — 7 days
Drug: Second period TWLO_C — Second Period: Single oral administration of 1 tablet of "Dong-a Bepotastine Besilate Tab"(Bepotastine Besilate 10mg)
  Other Names: "Dong-a Bepotastine Besilate Tab"
  Arms: TWLO → TWLO_C
Drug: Second period TWLO — Second Period: Single oral administration of 1 tablet of "Twolion Tab"(Bepotastine Besilate 10mg)
  Other Names: "Twolion Tab"
  Arms: TWLO_C → TWLO

SUMMARY:
An Open-Label, Randomized, 2-sequence, 2-period, Fasted Condition, Single-dose, Per Oral, Cross-over Study to Evaluate the Bioequivalence of "Dong-a Bepotastine Besilate Tab" (Bepotastine Besilate 10mg) and "Twolion Tab" (Bepotastine Besilate 10mg) in Healthy Volunteers

DETAILED DESCRIPTION:
1. Study design: An open-Label, randomized, 2-sequence, 2-period, fasted condition, single-dose, per oral, cross-over study
2. Administration method:

   The subject should maintain a minimum of 10 hours of empty stomach before administration, and give an oral dose of 1 tablets (Bepotastine Besilate 10 mg) with 150 mL of water at around 8 a.m. on the day of the test at room temperature. The test subject should not chew the drug or break it, but should swallow in whole with water. The difference in administration time between the test subjects is about one minute apart, considering the collection time.
3. Wash out period: 7 days
4. Blood collection time: Before the administration, 0.25, 0.5, 0.75, 1, 1.33, 1.67, 2, 3, 4, 6, 8, 12 hr after the administration (total 13 times)
5. Analysis: Measurement of the concentration of an unchangeable substance of Bepotastine in plasma

ELIGIBILITY:
Inclusion Criteria:

1. A person who aged 19 or older at the time of screening
2. No congenital or chronic diseases or pathological symptoms on screening
3. A person who is judged to be suitable for the study by the investigator based on the clinical laboratory examination
4. BMI of 18 to 30 (BMI calculation: kg/m2)
5. No history of gastrointestinal resection that may affect the absorption of drugs
6. No medical history of mental illness within five years prior to screening
7. A person who has fully understood the contents of the consent form for the study and signed the consent form voluntarily and recorded the date of signature
8. A person who is willing and able to follow all scheduled hospitalization and outpatient visits, medications, clinical laboratory examination and the terms of compliance
9. Female patients who were confirmed to be not pregnant at medical examination

Exclusion Criteria:

1. A person who has taken a drug that significantly induces (e.g., barbital) or inhibits the drug metabolic enzyme within 30 days prior to screening
2. A person who uses drugs that can affect the study within 10 days before screening
3. A person who is considered unsuitable to participate in the study by the investigator
4. A person who has participated in other clinical trials within three months prior to the first administration of the IP
5. A person who has had whole blood transfusion within 2 months or the apheresis within 2 weeks before screening
6. A person who is hypersensitive to venipuncture
7. A person with a history of regular alcohol intake within six months prior to screening:

   * Women: More than 14 cups/week
   * Men: More than 21 glasses/week (1 shot: 50 ml of soju, 30 ml of spirits, 250 ml of beer)
8. Hypersensitive to any of the IP components
9. Blood AST (GOT) or ALT (GPT) levels exceed the upper reference range limit by 2 times or γ-GTP levels exceed the upper reference range limit by 1.5 times
10. Lactating women
11. A person who does not agree to exclude the possibility of pregnancy using the contraception from the date of the first administration of the IP until the 7th day after the last administration.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Area Under the plasma Concetration versus time curve(AUClast) of Bepotastine Besilate | Before administration ~ 12 hours
Peak Plasma Concentration(Cmax) of Bepotastine Besilate | Before administration ~ 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea